CLINICAL TRIAL: NCT06497062
Title: Risk-stratified Treatment of Sonrotoclax Combined With Chemotherapy in Patients With Newly Diagnosed Acute Myeloid Leukemia: a Multicenter, Phase II Study
Brief Title: Phase II Study of Sonrotoclax Combined With Chemotherapy in the Treatment of Newly Diagnosed Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital (Other); BeiGene (Industry)
Responsible Party: Principal Investigator, Junmin Li, Head of hematology, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-2001-IIT
Record Dates: First submitted 2024-06-25; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Sonrotoclax; Risk-stratified; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Daunorubicin; Cytarabine; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Experimental: Sonrotoclax combined with intensive chemotherapy. Subjects receive induction therapy consisting of sonrotoclax combined with a 3+7 regimen. According to the ELN risks and MRD status, subjects who achieve composite complete remission (CRc) proceed with consolidation therapy, and allogeneic hematopoietic stem-cell transplant (allo-HSCT) can be included per investigator's decision.
  After the consolidation, subjects will receive sonrotoclax combined with azacitidine (AZA) alternating with AZA monotherapy every 2 cycles as maintenance therapy until intolerable toxicity, 12 months, relapse, death, withdrawal of informed consent, or study termination determined by investigators, whichever occurs first.
  Interventions: Drug: sonrotoclax; Drug: idarubicin/daunorubicin; Drug: Cytarabine; Drug: Azacitidine; Procedure: allo-HSCT

INTERVENTIONS:
Drug: sonrotoclax — Orally once daily, on D5-14. A 4-day dose ramp-up is required for the first induction. The dosing regimen will be determined in the Safety Run-in phase.
  If a second induction is needed, dose ramp-up is not required. In the consolidation therapy phase, subjects in the group with favorable risk and MRD negative do not need to receive Sonrotoclax treatment, and subjects in the group with favorable risk and MRD positive, or with intermediate and adverse risk will receive sonrotoclax on D1-7 at the target dose determined in the safety run-in phase, dose ramp-up is not required.
  In the maintenance therapy phase, subjects will receive once daily sonrotoclax on D1-14 at the target dose determined in the safety run-in phase.
  Other Names: BGB11417
Drug: idarubicin/daunorubicin — idarubicin: On D1-3, intravenously, 10 mg/m^2 for subjects aged <60 years, 6 mg/m^2 for subjects aged ≥60 years daunorubicin: On D1-3, intravenously, 60 mg/m^2 for subjects aged <60 years, 40 mg/m^2 for subjects aged ≥60 years
  Other Names: IDA/DNR
Drug: Cytarabine — In induction therapy phase: intravenously, 100 mg/m^2 on D1-7. In consolidation therapy phase: subjects with favorable-risk and MRD negative will receive cytarabine intravenously at 2 g/m^2/q12h for those aged <60 years, at 1g/m^2/q12h for those ≥60 years on D1-3 or 3+7 regimen, and subjects with favorable-risk and MRD positive or intermediate or adverse-risk will receive cytarabine intravenously at 1 g/m^2/d q12h on D1-3(in combination with sonrotoclax).
  Other Names: Ara-c
Drug: Azacitidine — 75 mg/m^2, subcutaneously, once daily, on D1-7
  Other Names: AZA
Procedure: allo-HSCT — Per standard of procedure

SUMMARY:
This single-armed study aims to investigate the safety and efficacy of sonrotoclax in combination with intensive chemotherapy in subjects with newly diagnosed AML. Subjects will be stratified based on the genetic risk classification of 2022 European LeukemiaNet (ELN) recommendations and MRD status to receive specific consolidation therapy after the induction therapy.

DETAILED DESCRIPTION:
47 subjects who meet the eligibility criteria will receive no more than 2 cycles (each cycle is 28 days) of induction therapy with sonrotoclax on day5-14 combined with the standard 3+7 intensive chemotherapy regimen (3+7 regimen) containing cytarabine, and daunorubicin or idarubicin. In cycle(C)1 of induction therapy, sonrotoclax will be administered orally once daily by a 4-day dose rump-up of 20mg on Day(D)5, 40mg on D6, 80mg on D7, and 160mg on D8-14. The first 6 subjects will be enrolled in a Safety Run-in period in C1 to assess tolerability and determine the final sonrotoclax regimen. Within 42 days or before the next cycle of therapy, if ≤1 of 6 subjects has dose-limiting toxicities (DLT), the study will be continued with the sonrotoclax dose regimen as above, and if ≥2 of 6 subjects have DLTs, the dose will be adjusted. Adjustment may include reducing the dose, shortening the duration of each cycle, or terminating the study, based on the DLTs' characteristics.

Subjects who achieve a composite complete remission (CRc) after induction therapy will receive further consolidation therapy, which regimen will be decided based on the ELN risk at diagnosis and MRD status detected by MFC after induction therapy.

After consolidation, subjects will receive once daily sonrotoclax orally combined with azacitidine (AZA) subcutaneously once daily alternating with AZA monotherapy every 2 cycles as maintenance therapy until unacceptable toxicity, 12 months, recurrence, death, withdrawal of informed consent, or study termination determined by investigators.

This single-armed study aims to investigate the safety and efficacy of a risk-stratified regimen of sonrotoclax in combination with intensive chemotherapy in subjects with newly diagnosed AML.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed untreated acute myeloid leukemia patients;
2. Age range from 18 to 75 years old;
3. The Eastern Cooperative oncology Group (ECOG) score is ≤ 2 points;
4. The following organ functional conditions must be met:

   * Liver function (bilirubin<2mg/dL, AST and/or ALT<3 x ULN)
   * Renal function (blood creatinine clearance rate ≥ 30 mL/min)
   * Cardiac function (left ventricular ejection fraction ≥ 50%)
5. If the age is ≥ 60 years old, the following conditions must be further met;

   * Charlson comorbidity index (CCI) ≤ 1
   * Activity of Daily Living Scale (ADL)>100
   * No cognitive impairment, Mini Mental State Examination (MMSE) ≥ 28
   * No impairment of living ability, Short Physical Performance Battery Protocol (SPPB) ≥ 9
6. Women with fertility must have a negative serum pregnancy test ≤ 7 days before the first administration. In addition, they must use efficient contraceptive methods before the first dose of study medication, during the study treatment period, and for ≥ 180 days after the last dose of study medication.
7. Non infertile males must use efficient contraceptive methods during the study treatment period and within ≥ 90 days after the last dose of the study medication. During this period, they are not allowed to donate sperm.
8. The patient fully understands this study, obtains an informed consent form (ICF) signed by the patient or their legal representative, and follows the research protocol and follow-up process.
9. The expected lifespan is greater than 12 weeks.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL)；
2. Malignant tumor in the past 2 years, except for cured localized skin cancer, superficial bladder cancer, cervical cancer or cancer in situ of breast cancer, and localized prostate cancer with Gleason score ≤ 6;
3. Uncontrolled concurrent diseases, including but not limited to: ongoing or active uncontrolled infections, cardiovascular or mental illnesses/social situations that may limit compliance with research requirements;
4. It is known that the subjects are positive for hepatitis B or hepatitis C infection, except those whose viral load cannot be detected within 3 months (Note: patients with HBcAb+but HBsAg - can only meet the condition if hepatitis B virus (HBV) DNA cannot be detected in the detection with sensitivity ≤ 20 IU/mL. In this case, patients should receive regular monitoring of HBV DNA and receive prophylactic antiviral drug treatment according to the central diagnosis and treatment routine; Patients with HCV antibody+are eligible only if they cannot detect HCV RNA and are willing to monitor HCV reactivation；
5. Receive any moderate or strong CYP3A4 inhibitor (7 days or 5 half-lives, whichever is longer) or moderate or strong CYP3A4 inducer (14 days or 5 half-lives, whichever is longer) treatment before the first use of Sonrotoclax；
6. Patients who are known to have hypersensitivity reactions to any component in the study protocol;
7. Known central nervous system involvement in AML;
8. Previously received organ, bone marrow, or peripheral blood organ transplantation；
9. Participate in another therapeutic clinical study simultaneously；
10. Pregnant or lactating women, or male and female patients planning to have children during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-09-04 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
EFS | 2-year
  event free survival rate

SECONDARY OUTCOMES:
Composite complete remission rate | Up to cycle 2 (each cycle is 28 days)
  Complete remission/complete remission with partial hematological recovery/complete remission with incomplete hematological recovery
The complete remission rate of MRD negative | Up to cycle 2 (each cycle is 28 days)
  The complete remission rate of MRD negative
RFS | Only for subjects who have achieved CR, CRh, or CRi; The time from the first attainment of eligible remission (CR, CRh, or CRi) after the start of treatment to the recording of disease recurrence or death, whichever occurs first. Up to 24 months
  relapse free survival rate
OS | up to 24 months
  overall survival rate
AE, SAE | up to 24 months
  Adverse event，Serious adverse events
Early mortality rate | Within 30 and 60 days after the first study medication
  Mortality within 30 days after first study medication and within 60 days after first study medication

OTHER OUTCOMES:
MRD and long-term survival | up to 24 months
  Evaluate the correlation with EFS and OS by grouping different remission states of MRD at the end of induction therapy and consolidation therapy
HSCT rate | up to 24 months
  HSCT rate and exploration of the association between HSCT and EFS and OS

CONTACTS AND LOCATIONS:
Overall Officials: Junmin Li, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Wu M, Jin Z, Yang L, Huang X, Li W, Zhu H, Wang W, Chen Q, Liu L, Chen Z, Wang S, Li J. Risk-stratified treatment of sonrotoclax with chemotherapy in newly diagnosed acute myeloid leukemia: a study protocol. Future Oncol. 2025 Apr;21(8):953-958. doi: 10.1080/14796694.2025.2469487. Epub 2025 Feb 26. PMID 40008672